CLINICAL TRIAL: NCT07085715
Title: Optimizing Pan-Viral Screening and Linkage to Treatment and Vaccination Among GBMSM and Trans Women in Spain, Including PrEP Users and Those Awaiting Access: An Online Self-Sampling Pilot Study
Brief Title: Pan-Viral Screening and Linkage to Care Among GBMSM and Trans Women in Spain
Acronym: PAN-TESTATE
Status: Not yet recruiting | Type: Observational
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Other Study IDs: PAN-TESTATE; 2024-9767 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2025-07-08; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: HIV; Hepatitis B; Hepatitis C
Keywords: Self-sampling; Screening
MeSH Terms: conditions — Hepatitis B; Hepatitis C | interventions — Seroconversion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Online self-sampling testing strategy to enhance pan-viral testing (HBV, HCV, HIV) — The TESTATE website (https://testate.org/) will be expanded to include the offer of free HBV/HCV/HIV self-sampling kit. Users will log in and complete a sociodemographic, behavioral and hepB vaccination survey, which will include the HCVMOSAIC questionnaire. Users identified at HCV risk will be sent a DBS collection kit by post to detect HCV RNA, HBsAg and HIV Ab. Participants will self-collect the DBS sample by finger prick at home and send them to the laboratory by post. The results will be delivered online. All participants who return samples will receive an acceptance survey by email.
  All participants recruited into the study will be provided with online information about the study and given the opportunity to ask questions and clarify queries to the field coordinator by email or phone.

SUMMARY:
The World Health Organization (WHO) aims to eliminate viral hepatitis as a public health threat by 2030, with major reductions in hepatitis B and C incidence and mortality. However, hepatitis C virus (HCV) transmission has increased among gay, bisexual, and other men who have sex with men (GBMSM), especially those living with HIV. Practices such as chemsex, particularly involving injection drug use, have contributed to this rise. Hepatitis B virus (HBV) also remains a public health challenge due to the potential for chronic infection and severe liver damage. Hepatitis D virus (HDV), which requires HBV co-infection, further complicates clinical management.

This study aims to design, implement, and evaluate an online self-sampling testing strategy to enhance pan-viral testing (HBV, HCV, HDV, HIV) and improve linkage to care among GBMSM and transgender women (TW) in Spain.

The intervention will involve self-collected dried blood spot (DBS) samples for testing HBV surface antigen (HBsAg), HIV antibodies, and HCV RNA. Individuals testing positive for HBsAg will undergo further testing for HBV DNA and HDV infection. Those lacking protective levels of HBV antibodies will be referred for vaccination or revaccination.

The study will also assess the number of HIV-positive individuals who acquired the infection while waiting for access to PrEP, identifying missed prevention opportunities.

This non-randomized, single-arm, prospective national study will recruit adult GBMSM and TW through PrEP services, dating apps, NGOs, social media, and community outreach. Participants will complete an online risk assessment (using the HCV-MOSAIC algorithm) and receive self-sampling kits with instructions, lancets, Whatman cards, and prepaid envelopes. Results will be provided online, and those testing positive will be linked to confirmatory diagnosis and care.

Outcomes include estimates of HIV, HBV, HCV, and HDV prevalence; effectiveness of linkage to care; acceptability and usability of the intervention; and validation of DBS for HBsAg detection.

This study will provide critical evidence on the effectiveness of online self-sampling strategies for viral hepatitis and HIV among GBMSM and TW, supporting Spain's public health goals for prevention, early diagnosis, and linkage to care.

DETAILED DESCRIPTION:
Background: The World Health Organization (WHO) aims to eliminate viral hepatitis as a public health threat by 2030, targeting significant reductions in incidence and mortality for hepatitis B and C. Despite these goals, hepatitis C virus (HCV) transmission and acute infection rates have risen among gay, bisexual, and other men who have sex with men (GBMSM), especially those with HIV. Chemsex, particularly involving drug injection, is a notable risk factor. Hepatitis B virus (HBV) also poses a significant public health challenge, with chronic hepatitis B leading to severe liver damage in a significant portion of those infected. Hepatitis D virus (HDV), which requires HBV co-infection, adds further complexity to the management of viral hepatitis. Integrating evidence-based interventions for HIV and STI prevention, including effective screening and linkage to care, is urgently needed.

Objectives: This study aims to design, implement, and evaluate an online self-sampling testing strategy to enhance pan-viral testing (HBV, HCV, HDV, HIV) and improve linkage to care among GBMSM and transgender women (TW) in Spain. Specific objectives include:

1. Designing and implementing an online self-sampling pilot intervention for HBV, HIV, and viremic HCV detection using dried blood spot (DBS) samples, and following up on positive HBV cases for HDV co-infection.
2. Analyzing the intervention's effectiveness in reaching and identifying undiagnosed infections among GBMSM and TW not recently tested for HIV and viral hepatitis.
3. Identifying individuals who have not vaccine-induced protective levels against HBV and linking them to vaccination (or revaccination) services.
4. Evaluating the intervention's acceptability among GBMSM and TW inSpain.
5. To identify the number of individuals with HIV infection while they are waiting PrEP (missed opportunities to prevent HIV infection) A secondary objective is to validate DBS samples for detecting HBV surface antigen (HBsAg).

Methods: This non-randomized single-arm prospective and national study will recruit adult GBMSM and TW through PrEP services, social media, gay dating apps, NGOs, and outreach interventions. Participants will complete a risk assessment using the HCV-MOSAIC algorithm, and eligible individuals will receive a self-sampling kit for HBV, HCV, and HIV testing. The kits will include instructions, a lancet, a Whatman card for DBS collection, and a pre-paid return envelope. Samples will be analyzed by a reference laboratory for HBsAg, HIV antibodies, and HCV RNA. Participants will receive their results online, with follow-up for those testing positive to confirm diagnoses and linkage to care. Those who test positive for HBsAg will be further tested for other tests, including HBV DNA, and HDV infection.

Expected Outcomes: The study will estimate HBV, HDV, HCV, and HIV prevalences, assess linkage to care and treatment outcomes, and evaluate the acceptability and usability of the self-sampling intervention. Additionally, the validation of DBS for HBsAg detection will provide crucial data for future screening strategies.

Conclusion: This study will provide valuable insights into the effectiveness of self-sampling interventions for viral hepatitis and HIV among GBMSM and TW, contributing to public health efforts to reduce the burden of these infections in Spain. To identify the number of individuals with HIV infection while they are waiting PrEP (missed opportunities to prevent HIV infection)

ELIGIBILITY:
Inclusion Criteria:

* Men self-reporting being gay, bisexual, and other men who have sex with men (GBMSM) or transgender women
* 18 years old or older
* Residing in Spain
* Accepting to participate and signing the informed consent
* Including those who are in PrEP or waiting access to PrEP; regardless of their HIV status (HIV-negative or HIV-positive), and considered at risk for HCV acute infection using the MOSAIC validated algorithm (score of 2 or higher).

Exclusion Criteria:

* <18 years old
* No GBMSM or transgender women
* Non-residents in Spain
* No signing the informed consent
* Not considered at risk for HCV acute infection using the MOSAIC validated algorithm (score lower than 2).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gay, bisexual, and other men who have sex with men (GBMSM) and transgender women residing in Spain
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reach and Identification of Undiagnosed HBV/HCV/HIV Infections | October 2025 - September 2026
  Number of GBMSM and TW reached by the intervention Number of undiagnosed HBV, HCV, and HIV infections identified among participants
Linkage to Care_1 | October 2025 - September 2026
  • Number and proportion of participants with positive results linked to appropriate care and follow-up.
Linkage to care_2 | October 2025 - September 2026
  • Follow-up and cure rates for HCV infection among participants with positive results.
Linkage to care_3 | October 2025 - September 2026
  • Number of individuals identified as not vaccinated against hepatitis B and linked to vaccination services.
Intervention Usability and Acceptability_1 | October 2025 - September 2026
  • Number of participants consulting their results.
Intervention Usability and Acceptability_2 | October 2025 - September 2026
  • Participant satisfaction with the intervention, perceived advantages and disadvantages, suggestions for improvement..
Intervention Usability and Acceptability_3 | October 2025 - September 2026
  • Percentage of participants repeating HIV/HBV/HCV screening.

SECONDARY OUTCOMES:
Effectiveness of DBS Screening_1 | October 2025 - September 2026
  Proportion of participants with confirmed positive results for HBV, HCV, and HIV using DBS self-samples.
Effectiveness of DBS Screening_2 | October 2025 - September 2026
  Validation metrics for DBS samples in detecting HBsAg, including the area under the ROC curve and the 95% confidence interval.
Missed Opportunities for HIV Prevention | October 2025 - September 2026
  • Number of participants on the waiting list for PrEP who are diagnosed with HIV.
Sociodemographic and Risk Behavior Analysis_1 | October 2025 - September 2026
  • Comparison of sociodemographic characteristics and risk behaviors between positive and negative participants.
Sociodemographic and Risk Behavior Analysis_2 | October 2025 - September 2026
  • Data disaggregated by gender, migratory status, and sexual orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Agusti, MSc, PhD, Study Director — ico oncologia

IPD SHARING:
Plan to Share IPD: No